CLINICAL TRIAL: NCT04732637
Title: Evaluating the Use of Flavour-stimulated Oral Fluids Collection for Severe Acute Respiratory Syndrome Coronavirus 2 Detection by Reverse Transcriptase Polymerase Chain Reaction and Enzyme Linked Immunosorbent Assay - a Concordance Study.
Brief Title: Concordance Between Buccal Cavity Swab and Nasopharyngeal Swab for SARS-CoV-2 (COVID-19) Detection by RT-PCR and ELISA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Datar Cancer Genetics Limited (Industry)
Collaborators: Test At Home Pte. Ltd (Unknown); National University of Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: U1111-1264-2742
Record Dates: First submitted 2021-01-28; First posted 2021-02-01 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Covid19
Keywords: COVID19; Nasopharyngeal Swab; Self Collection; Chewable; Lollipop
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biological samples collected via nasopharyngeal swaps and 'lollipop' buccal mucosa swabs and used for extraction of viral nucleic acids
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID Positive: Individuals who have recently tested positive for COVID19 by RTPCR, with active infection.
  Interventions: Diagnostic Test: Test At Home's Proprietary "Lollipop" Buccal Cavity Swab
- COVID Negative: Individuals who have recently tested negative for COVID19 by RTPCR.
  Interventions: Diagnostic Test: Test At Home's Proprietary "Lollipop" Buccal Cavity Swab

INTERVENTIONS:
Diagnostic Test: Test At Home's Proprietary "Lollipop" Buccal Cavity Swab — Self-collected Test At Home's proprietary "Lollipop" Buccal Cavity Swab with VTM.
  Other Names: Self Collection Buccal Cavity Swab; Buccal Cavity Swab

SUMMARY:
Nasopharyngeal Swabs (NPS) used to test for Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) infection can cause mild to severe discomfort in addition to increasing the risk of transmission. The present study evaluates Test At Home's proprietary self-collection method based on a chewable buccal cavity swab ("lollipop") that stimulates oral fluid collection. The novel method is compared against a contemporary nasal swab collected by a qualified healthcare worker.

DETAILED DESCRIPTION:
Nasopharyngeal Swabs (NPS) are used to test for Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) infection. For this, a swab is inserted deep into the back of the nose to collect a sample. It can cause discomfort for most people. It also increases the risk of transmission and other challenges. The present study aims to develop a more convenient method of collecting samples for COVID-19 testing. The study is based on the hypothesis that saliva collection using the proprietary flavour-stimulated 'Lollipop' swab (LPS) can be a more viable alternative to NPS.

The study aims to establish the comparative efficacy of SARS-Cov-2 infection assessment using Test At Home's proprietary "lollipop" buccal cavity swab (LPS) that simulates oral fluid collection via flavouring and mastication (self-collection) using the contemporary nasal swab collection (by health worker) as standard.

For the present study, 300 pairs of matched nasopharyngeal swab (NPS) (health care worker collected) and simulated oral fluid specimens (self-collected) will be obtained from 150 Coronavirus Disease -19 (COVID-19) positive patients and 150 COVID 19 negative individuals.

Test Method 1: Self-collected Test At Home's proprietary "lollipop" buccal cavity swab with Viral Transport Medium (VTM) will be evaluated using the Standard 'TaqPath™' COVID-19 Conformité Européenne - In Vitro Diagnostic (CE-IVD) Reverse Transcriptase-Polymerase Chain Reaction (RT-PCR) which is approved by the Indian Council of Medical Research (ICMR)

Test Method 2: Self-collected Test At Home's proprietary "lollipop" buccal cavity swab with VTM will be evaluated using National University of Singapore (NUS) developed Enzyme Linked Immunosorbent Assay (ELISA) Method.

Active Comparator : Health worker collected Nasopharyngeal Swab (NPS) with VTM which will be evaluated using the Standard TaqPath™ COVID-19 CE-IVD RT-PCR which is approved by the Indian Council of Medical Research (ICMR).

The diagnostic performance of using NPS and Oral fluids will be statistically compared to determine concordance of positive and negative findings and establish the performance characteristics of the Test Methods.

ELIGIBILITY:
Inclusion Criteria:

1. Males and Females
2. Adults
3. Known COVID-19 positive by RTPCR (with active infection) OR Known COVID-19 negative by RTPCR (tested within 7 days)
4. Provision of Informed Consent
5. Willing to provide Nasopharyngeal Swab as well as Buccal Cavity Swab

Exclusion Criteria:

1. Pediatric patients.
2. Inability to provide Informed Consent.
3. Inability to provide Nasopharyngeal Swab and / or Buccal Cavity Swab.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult males and females, who have understood the aims, scope, benefits and risks of the study as well as study procedures and provide Informed Consent are eligible to participate. The Study will recruit one hundred and fifty (150) individuals who are known COVID-19 positive (confirmed by RTPCR) and have active infection. The Study will also recruit one hundred and fifty (150) individuals who are known COVID-19 negative (confirmed by RTPCR within the last 7 days).
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-03-31 (Estimated); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Concordance between buccal cavity swab and contemporary nasal swab. | Baseline / Day 0 (At first collection)
  Three-way concordance of SARS-Cov-2 infection assessment between Test At Home's "Lollipop" buccal cavity swab (assessed by RTPCR and ELISA) and contemporary nasal swab (assessed by RTPCR).

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Manoharan, PhD, Principal Investigator — Test At Home Pte. Ltd., Singapore - India.; Paul Macary, PhD, Principal Investigator — National University of Singapore; Saket Jhajharia, PhD, Principal Investigator — Test At Home Pte. Ltd., Singapore - India; Terence Tan, MBBS, Principal Investigator — Test At Home Pte. Ltd., Singapore - India.; Vineet Datta, MD, Principal Investigator — Datar Cancer Genetics Limited, United Kingdom - India; Kanupriya Batra, MBA, Principal Investigator — Test At Home Pte. Ltd., Singapore - India.
Locations (1):
- Datar Cancer Genetics, Nashik, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided
Individual Participant Data (IPD) may be made available to qualified researchers upon written request with declaration of intent to use and after signing of a Confidentiality Agreement / Non Disclosure Agreement (NDA).